CLINICAL TRIAL: NCT03820674
Title: A Telerehabilitation Intervention to Reduce the Impact of Fatigue in People With Congestive Heart Failure and Chronic Fatigue
Brief Title: A Telerehabilitation Intervention for People With Heart Failure and Chronic Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Carolina University (Other)
Responsible Party: Principal Investigator, Young Joo Kim, Assistant Professor, East Carolina University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UMCIRB 16-000078
Record Dates: First submitted 2019-01-24; First posted 2019-01-29 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Heart Failure
Keywords: Heart Failure; Fatigue; Rehabilitation; Occupational Therapy
MeSH Terms: conditions — Heart Failure; Fatigue

STUDY DESIGN:
Intervention Model Description: Both groups received 6-week interventions.
Who Masked: Participant
Masking Description: Participants are blinded to their group assignment. Assessors and interventionists were not blinded to the group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Energy Conservation plus Problem Solving Therapy Intervention (Experimental): Receiving experimental intervention
  Interventions: Other: Energy Conservation plus Problem Solving Therapy
- Health Education Intervention (Active Comparator): Receiving control intervention
  Interventions: Other: Health Education Intervention

INTERVENTIONS:
Other: Energy Conservation plus Problem Solving Therapy — EC-PST is a client-centered intervention aiming to guide people with chronic fatigue to create their own solutions so that they can generalize those learned solutions and strategies to other fatigue-related problems even after completing the study participation. Some of the topics covered during the first two introductory sessions are facts regarding fatigue, budgeting and banking energy, and the introduction of EC+PST Intervention.
  Arms: Energy Conservation plus Problem Solving Therapy Intervention
Other: Health Education Intervention — The interventionist will be the PI, an occupational therapist (co-I), or OT graduate student who will be trained in the health education topics. During the Health Education sessions, participants will be educated on health-related topics relevant to CHF and EC strategies, although they will not learn how to apply the information to their daily life. Health Education Workbook containing information on the topics taught during the sessions will be provided during the Pretest visit and used throughout the Health Education sessions.
  Arms: Health Education Intervention

SUMMARY:
This study compares the effectiveness of a 6-week Energy Conservation + Problem Solving Therapy Intervention to Health Education Intervention for reducing the fatigue impact and fatigue level and improving the level of participation in instrumental, leisure, and social activities in people with heart failure associated fatigue. Half of the participants received Energy Conservation + Problem Solving Therapy Intervention, and the other half received Health Education Intervention.

DETAILED DESCRIPTION:
Energy Conservation+Problem Solving Therapy (EC+PST) Intervention: In this study, the EC+PST Intervention will ideally occur twice a week for 6 weeks with each session lasting approximately 30 minutes. The intervention will be individually delivered via telehealth; therefore, participants will receive the intervention in their home to minimize fatigue from the intervention.

Health Education Intervention: The Health Education Intervention will occur once a week for 6 weeks with each session lasting approximately 30 minutes. The Health Education Intervention will be delivered via telehealth; therefore, participants will receive the intervention at their convenient quiet place to minimize fatigue from the intervention.

ELIGIBILITY:
Inclusion Criteria:

(a) a minimum 6 months since diagnosed with HF and 3 months post-hospitalization, (b) reporting of moderate to severe fatigue by scoring ≥4 according to Fatigue Severity Scale, (c) living in the community, (d) having access to the internet or telephone in the place of residence, (e) having functional English fluency, and (f) having functional vision to operate the tablet computer.

Exclusion Criteria:

1. had a score of ≥9 in Short Blessed Test indicating cognitive impairment
2. were classified as having New York Heart Association (NYHA) Functional Classification level IV on their medical record

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-06-17 (Actual); Primary Completion 2018-05-02 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Changes in Fatigue Impact Scale (FIS) | Pretest (Week 0), Posttest (Week 7)
  The FIS is a 40-item measure that assesses the impact of fatigue on daily life in three different dimensions: Cognitive (10 items), Physical (10 items), and Psychosocial functioning (20 items). Each item is rated on a 5-point scale ranging from 0 (no problem) to 4 (extreme problem), and the global score is the sum of 40 items, ranging from 0 to 160.
Changes in Patient-Reported Outcomes Measurement Information System (PROMIS) - Short Form Ver 1.0 Fatigue 8a | Pretest (Week 0), Posttest (Week 7)
  The PROMIS Fatigue 8a is a test measuring the experience and impact of fatigue. This assessment consists of 8 questions on fatigue experience and impact, and the raw score is converted to T-score (50% is the mean of the population). Higher the T-score, worse the fatigue.
Changes in Activity Card Sort (ACS) | Pretest (Week 0), Posttest (Week 7)
  The ACS is a measure of the participation level in instrumental, leisure, and social activities. The ACS uses 89 photographs to calculate the percentage of retained activities since their diagnosis

REFERENCES:
- [Derived] Kim YJ, Radloff JC, Crane PA, Bolin LP. Rehabilitation Intervention for Individuals With Heart Failure and Fatigue to Reduce Fatigue Impact: A Feasibility Study. Ann Rehabil Med. 2019 Dec;43(6):686-699. doi: 10.5535/arm.2019.43.6.686. Epub 2019 Dec 31. PMID 31918531